CLINICAL TRIAL: NCT03234348
Title: MAGnesium-based Bioresorbable Scaffold and Vasomotor Function in Patients With Acute ST Segment Elevation Myocardial Infarction
Brief Title: MAGnesium-based Bioresorbable Scaffold in ST Segment Elevation Myocardial Infarction
Acronym: MAGSTEMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Manel Sabate, MD, MD, PhD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAG-01
Record Dates: First submitted 2017-07-24; First posted 2017-07-31 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Acute Coronary Syndrome; ST Segment Elevation Myocardial Infarction; Stent
Keywords: biodegradable stent; STEMI; Magnesium bioresorbable; Vasomotion
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to one of two groups:
  MAGMARIS stent arm or ORSIRO stent arm in the ratio of 1:1
Who Masked: Participant, Outcomes Assessor
Masking Description: Neither the participant ot the outcomes assessor will be aware of the treatment received. The patient will be blinded until the primary endpoint is reached (1 year follow-up).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magmaris (Experimental): Percutaneous coronary intervention by means of Magnesium-based sirolimus-eluting bioresorbable scaffold implantation after proper lesion preparation by balloon predilatation and/or manual thrombectomy.
  Interventions: Device: Percutaneous coronary intervention
- Orsiro (Placebo Comparator): Percutaneous coronary intervention by means of Biodegradable polymer sirolimus-eluting stent implantation after proper lesion preparation by balloon predilatation and/or manual thrombectomy.
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — PCI + stent implantation
  Other Names: stent implantation

SUMMARY:
This is a prospective, randomized, active control, single-blind, non-inferiority, multicenter clinical trial. 148 subjects will be registered at up to 10 Spanish sites. Subjects will be followed for 5 years.

All eligible patients (STEMI < 12 hours from onset of chest pain) will be randomized to

* Biotronik MAGMARISTM Sirolimus Eluting Bioresorbable Vascular Scaffold System (M-BRS) or
* Biotronik ORSIRO Sirolimus Eluting Coronary Stent System

Endothelium-independent vasomotor response (NTG injection) will be analyzed at 12 months angiographic follow-up (Primary endpoint).

In a subgroup of 40 patients Optical Coherence Tomography will be performed after the procedure and at 12 months follow-up.

Angiographic (QCA pre- and post-procedure and at 12 months follow-up), OCT data (at 12 months follow-up) will be analyzed off-line by an independent core lab.

ELIGIBILITY:
Inclusion Criteria:

Clinical:

1. At least 18 years of age.
2. ST-segment elevation Myocardial Infarction documented in an ambulance or in a Cathlab, with ≥2 mm ST segment elevation in at least two contiguous leads, presenting in the Cathlab <12 hours after the onset of symptoms lasting ≥20 min requiring primary PCI.
3. Target lesion must be a de-novo lesion located in a native vessel.
4. The patient accepts Informed Consent
5. The patient understands and accepts clinical follow-up and angiographic control.

   Angiographic:
6. Vessel size should match available M-BRS scaffold sizes (≥2.75 mm, and ≤3.7 mm by visual assessment).
7. Lesion preparation by either manual thrombectomy or pre-dilatation has been successful, with opening of the vessel and TIMI ≥2 and residual stenosis <20%.

Exclusion Criteria:

1. Pregnancy.
2. Known intolerance to aspirin, heparin, stainless steel, sirolimus, and contrast material.
3. Distal vessel occlusion after recanalization
4. STEMI due to stent/scaffold thrombosis
5. Severe tortuous, calcified or angulated coronary anatomy of the study vessel that in the opinion of the investigator would result in sub-optimal m-BRS placement.
6. Fibrinolysis prior to PCI
7. Known thrombocytopenia (PLT< 100,000/mm3)
8. Active bleeding or coagulopathy or patients at chronic anticoagulation therapy
9. Cardiogenic Shock
10. Significant comorbidities precluding clinical/angiographic FU (as judged by investigators)
11. Major planned surgery that requires discontinuation of dual antiplatelet therapy.
12. Diffuse coronary artery disease that will require CABG
13. Chronic kidney disease with GFR<30 ml/min

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
In-stent/scaffold vasodilatory endothelium independent response | 12 months follow-up
  in-stent/scaffold vasodilatory response ≥3% (delta in mean lumen diameter) after nitroglycerin injection

SECONDARY OUTCOMES:
Device success | Immediate after the procedure
  implantation of the intended device with attainment of <30% residual stenosis of the target lesion and TIMI ≥2
Procedure success | Up to 7 days
  device success and no in-hospital cardiac events: death, repeat MI, TVR or stent/scaffold thrombosis
Device-oriented Composite Endpoint (DOCE) | 1, 6 months, 1,2,3,4,5 years
  Combined of cardiac death, Target vessel MI, or clinically-indicated target lesion revascularization
Cardiac death | 1, 6 months, 1,2,3,4,5 years
  ARC definition
Target vessel MI | 1, 6 months, 1,2,3,4,5 years
  ARC definition
Clinically driven target lesion revascularization | 1, 6 months, 1,2,3,4,5 years
  ARC definition-Ischemia driven revascularization
Stent/scaffold thrombosis | 1, 6 months, 1,2,3,4,5 years
  ARC definition: definite, probable, possible, acute, subacute, late and very late
Patient oriented endpoint (POCE) | 1, 6 months, 1,2,3,4,5 years
  Combined of all-cause death, any repeat myocardial infarction and any revascularization
All-cause death | 1, 6 months, 1,2,3,4,5 years
  All-cause death rate
Any repeat myocardial infarction | 1, 6 months, 1,2,3,4,5 years
  According to WHO extended definition
Any revascularization | 1, 6 months, 1,2,3,4,5 years
  Any repeat intervention in the patient
Target lesion revascularization | 1, 6 months, 1,2,3,4,5 years
  ARC definition
Target vessel revascularization | 1, 6 months, 1,2,3,4,5 years
  ARC definition
MLD | Baseline and 1 year follow-up
  Minimal lumen diameter by QCA
%DS | Baseline and 1 year follow-up
  percentage diameter stenosis by QCA
Acute gain | Baseline
  MLD post - MLD pre by QCA
Late loss | 1 year
  MLD post - MLD at 1 year follow-up by QCA
Binary restenosis | 1 year
  % of patients with >50% DS at 1 year follow-up by QCA
Lumen area | 1 year follow-up
  Mean and minimum lumen area of the stented/scaffolded segment by OCT
Mean lumen volume | 1 year follow-up
  mean lumen volume of the stented/scaffolded segment by OCT
% strut malapposition | 1 year follow-up
  mean area of strut malapposition by OCT
Tissue Prolapse | 1 year follow-up
  presence and % of lumen area occupied by tissue prolapse by OCT
Neointimal hyperplasia | 1 year follow-up
  mean intra-stent/scaffold area occupied by neointimal hyperplasia by OCT
Healing index | 1 year follow-up
  Index obtained by a combination of % malapposition, % coverage, % tissue prolapse by OCT
Strut coverage | 1 year follow-up
  Presence and amount of tissue covering the strut of the stent/scaffold by OCT
RUTTS | 1 year follow-up
  Ratio of Uncovered to Total Stent/scaffold Struts Per Cross Section (RUTTS) score of ≤30% of the target stent/scaffold as determined by OCT pullback
in-stent/in-scaffold endothelium-dependent vasomotion | at 12 months
  % change in mean luminal dimeter on the treated segment after acetylcholine infusion

CONTACTS AND LOCATIONS:
Overall Officials: Manel Sabaté, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (11):
- Spain (11):
  - Hospital General de Alicante, Alicante
  - Hospital Clínic, Barcelona
  - Hospital Sant Pau, Barcelona
  - Hospital Universitari Bellvitge, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Clínico San Carlos, Madrid
  - Hospital La Princesa, Madrid
  - Hospital Puerta de Hierro Majadahonda, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Alvaro Cunqueiro, Vigo

IPD SHARING:
Plan to Share IPD: Yes
Data on primary/secondary outcomes on individual basis may be shared with other researchers once main report as been published and review and approval of the research proposal by the steering committee of the Magstemi Trial
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data on primary/secondary outcomes on individual basis may be shared with other researchers once main report as been published and review and approval of the research proposal by the steering committee of the Magstemi Trial

REFERENCES:
- [Background] Brugaletta S, Cequier A, Alfonso F, Iniguez A, Romani S, Serra A, Salinas P, Goicolea J, Bordes P, Del Blanco BG, Hernandez-Antolin R, Pernigotti A, Gomez-Lara J, Sabate M. MAGnesium-based bioresorbable scaffold and vasomotor function in patients with acute ST segment elevation myocardial infarction: The MAGSTEMI trial: Rationale and design. Catheter Cardiovasc Interv. 2019 Jan 1;93(1):64-70. doi: 10.1002/ccd.27825. Epub 2018 Sep 9. PMID 30196572
- [Result] Sabate M, Alfonso F, Cequier A, Romani S, Bordes P, Serra A, Iniguez A, Salinas P, Garcia Del Blanco B, Goicolea J, Hernandez-Antolin R, Cuesta J, Gomez-Hospital JA, Ortega-Paz L, Gomez-Lara J, Brugaletta S. Magnesium-Based Resorbable Scaffold Versus Permanent Metallic Sirolimus-Eluting Stent in Patients With ST-Segment Elevation Myocardial Infarction: The MAGSTEMI Randomized Clinical Trial. Circulation. 2019 Dec 3;140(23):1904-1916. doi: 10.1161/CIRCULATIONAHA.119.043467. Epub 2019 Sep 25. PMID 31553204
- [Derived] Gomez-Lara J, Ortega-Paz L, Brugaletta S, Cuesta J, Romani S, Serra A, Salinas P, Garcia Del Blanco B, Goicolea J, Hernandez-Antolin R, Antuna P, Romaguera R, Regueiro A, Rivero F, Cequier A, Alfonso F, Gomez-Hospital JA, Sabate M; Collaborators. Bioresorbable scaffolds versus permanent sirolimus-eluting stents in patients with ST-segment elevation myocardial infarction: vascular healing outcomes from the MAGSTEMI trial. EuroIntervention. 2020 Dec 4;16(11):e913-e921. doi: 10.4244/EIJ-D-20-00198. PMID 32310130